CLINICAL TRIAL: NCT07339514
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study of ER2001 Intravenous Injection in Adults With Early Manifest Huntington's Disease.
Brief Title: A Phase I Clinical Study of ER2001 Injection for the Treatment of Early Manifest Huntington's Disease.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ExoRNA Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ER2001-102; CTR20243121 (Registry Identifier: the Study Number on chinese website(http://www.chinadrugtrials.org.cn))
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: Biological Product.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1.ER2001 - 0.08mg/kg (Active Comparator): The planned duration of the treatment is 6 weeks, and ER2001 will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.
  Interventions: Drug: ER2001 intravenous injection
- 2.ER2001 - 0.32mg/kg (Active Comparator): The planned duration of the treatment is 6 weeks, and ER2001 will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.
  Interventions: Drug: ER2001 intravenous injection
- 3.Placebo Intravenous Injection (Placebo Comparator): The planned duration of the treatment is 6 weeks, and Placebo will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ER2001 intravenous injection — The drug dose is 0.08mg/kg, or 0.32mg/kg. The planned duration of each patient's treatment is 6 weeks, and ER2001 will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.
  Arms: 1.ER2001 - 0.08mg/kg; 2.ER2001 - 0.32mg/kg
Drug: Placebo — Placebo Injection, The planned duration of the treatment is 6 weeks, and Placebo will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.
  Arms: 3.Placebo Intravenous Injection

SUMMARY:
This is a dose escalation and expansion clinical study to evaluate the safety, tolerability, PK profile and preliminary efficacy of ER2001 Injection vs. placebo in subjects with definitive diagnosis of early manifest HD.

The study consists of a dose escalation phase (Part A, an open-label without placebo, which will be carried out firstly) and a dose expansion phase (Part B,randomized, blinded, placebo-controlled), both of which include a screening period (4 week prior to the first administration), a treatment period (for 6 consecutive weeks, once a week [QW] for 6 weeks), and a safety follow-up period (24 weeks).

DETAILED DESCRIPTION:
Two dose levels will be included in the dose escalation phase, and subjects will be in cohorts (Cohort 1, and Cohort 2) in sequence to receive the investigational drug. Either 3 or 6 subjects will be enrolled in each cohort. Dose escalation from the current cohort to the next cohort will be determined through joint review by the sponsor and the IDMC, typically based on the number of DLT(dose-limiting toxicity)s observed in subjects. If one DLT occurs in a cohort, additional 3 subjects will be enrolled in that cohort, with a total of 6 subjects. If one DLT occurs in the low-dose cohort while the administration is ongoing in the high-dose cohort, recruitment of subjects in the high-dose cohort should be held until all enrolled subjects have completed their dosing regimen and a safety assessment of at least 7 days after completion of the treatment. In addition, the IDMC will hold a meeting to decide whether further actions are necessary, e.g., dose interruption or reduction for subjects in the high-dose cohort. If two DLTs occur in a cohort, the dose will be discontinued in that cohort and any active higher dose cohorts. No more than one subject within the same cohort should initiate the treatment on the same day.

Based on review of safety, tolerability, PK and exploratory PD results in the dose escalation phase, dose expansion will be performed in 1 or 2 cohort(s) at the recommended dose levels. For the dose expansion phase, 9 subjects (including 3 subjects in the placebo control group) will be enrolled for each dose level cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has documented ability to understand the written study informed consent forms (ICFs) at the time of screening and has provided signed written informed consent prior to any study procedures.

2.25 Years to 55 Years. Gender is not limited. 3.Early manifest HD as defined by a UHDRS total functional capacity (TFC) score of 10 to 13 and a diagnostic classification level (DCL) of 4.

4.HTT gene expansion testing with the presence of ≥40 CAG repeats. 5.Ability to undergo and tolerate MRI scans. 6.Ability to undergo and tolerate lumbar puncture. 7.All HD medications given for motor, behavioral, and cognitive symptoms have been stable for 3 months prior to Screening.

8.Other concomitant medications have been stable for 1 month prior to Screening.

9.organ function measured prior to administration of study treatment. 10.Postmenopausal or evidence of non-childbearing status for women of childbearing potential. Male patients must use a condom during treatment and for 6 months after the last dose of ER2001 when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

1. History of attempted suicide or suicidal ideation with plan (i.e., active suicidal ideation) that required hospital visit and/or change in level of care within 12 months prior to screening.
2. Current active psychosis, confusional state, or violent behavior.
3. Bleeding tendency or history of coagulation disorder; As long as the investigator confirms that there is no evidence of bleeding tendency or coagulation dysfunction at present.
4. ECG with corrected QT interval (QTc) > 450 ms and/or indication of uncontrolled cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction,congestive heart failure, electrolyte disturbances, etc.)
5. Patients with HIV, Treponema pallidum, Hepatitis B, or Hepatitis C infection.
6. Need to take antiretroviral drugs, including antiretroviral drugs as preventive treatment.
7. Current or recurrent disease, infection, or other significant concurrent medical condition or medications that could confound clinical and laboratory evaluations or could affect a subject's safety or their ability to undergo the neurosurgical procedure or comply with the procedures and study visit schedule.
8. Clinical diagnosis of chronic migraines.
9. Presence of an implanted deep brain stimulation device, ventriculoperitoneal or other CSF shunt, or other implanted catheter.
10. Preexisting structural brain lesions (such as tumor, arteriovenous malformation) as assessed by a centrally read MRI scan during the screening period.
11. Any history of gene therapy, RNA or DNA investigational agents, such as antisense oligonucleotides (ASO), cell transplantation or any other experimental brain surgery.
12. Treatment with investigational therapy within 4 weeks prior to screening or 5 drug elimination half-lives of investigational therapy, whichever is longer.
13. Unable or unsafe to perform lumbar puncture on the patient.
14. In the Investigator's judgment, that Parkinson's disease, multiple system atrophy and other dystonia diseases may be combined.
15. Patients who are hypersensitive to any ingredients in the formulation of ER2001.
16. Malignancy within 5 years of screening, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
17. Concurrent or planned concurrent participation in any interventional clinical study, including explicit pharmacological and non- pharmacological interventions. Observational studies are acceptable.
18. Any serious medical condition or clinically significant laboratory, vital signs, or abnormalities at screening that, in the Investigator's judgment, precludes the patient's safe participation in and completion of the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of adverse events (AEs) and serious adverse events (SAEs). | Approximately 7.5 months
  To evaluate the safety and tolerability of ER2001 injection or placebo.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Approximately 7.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.
Terminal half-life (t1/2) | Approximately 7.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.
Area under the plasma concentration versus time curve from time 0 to the last quantifiable concentration (AUC0-t). | Approximately 7.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.
Maximum concentration (Cmax) in cerebrospinal fluid (CSF) | Approximately 7.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.

OTHER OUTCOMES:
Change from baseline in the concentration of mutant huntingtin (mHTT) protein in cerebrospinal fluid (CSF) | Approximately 7.5 months
  To assess the dose-response relationship of ER2001 injection on mHTT protein change from baseline in cerebrospinal fluid (CSF).
Immunogenicity | Approximately 7.5 months
  To collect the incidence of Anti-Drug Antibodies (ADAs).
change in multicytokine levels from baseline | Approximately 7.5 months
  To evaluate the effect of ER2001 injection on changes in multiple cytokine levels in patients with Huntington's disease
Change from baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity (TFC) score | Approximately 7.5 months
  UHDRS is a research tool developed by Huntington Disease (HD) Study Group to provide a uniform assessment of the clinical features and course of HD. The UHDRS TFC comprises 5 functional domains associated with disability (occupation, finances, domestic chores, activities of daily living, and care level), with scores on each item ranging from 0 to either 2 or 3. The TFC total score is the sum of the 5 TFC items and can range from 0 to 13, with greater scores indicating higher functioning. Negative change from baseline indicates worsening.
Change from baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score (TMS) score | Approximately 7.5 months
  UHDRS is a research tool developed by Huntington Disease (HD) Study Group to provide a uniform assessment of the clinical features and course of HD. The UHDRS TMS assesses all the motor features of HD and includes maximal chorea, maximal dystonia, ocular pursuit, saccade initiation and velocity, dysarthria, tongue protrusion, finger tapping, hand pronation and supination, luria, rigidity, bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these was rated on a scale of 0 (normal motor function) to 4 (severely impaired motor function). TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function). Lower TMS scores indicate better motor function.

CONTACTS AND LOCATIONS:
Overall Officials: jinsheng zeng, Ph.D, Study Chair — First Affiliated Hospital of Sun Yat-sen University; pingyi xu, Ph.D, Principal Investigator — First Affiliated Hospital of Guangzhou Medical University; huifang shang, Ph.D, Principal Investigator — West China Hospital
Locations (3):
- China (3):
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - West China Hospital of Sichuan University, Chengdu, Sichuan